CLINICAL TRIAL: NCT00114140
Title: A Phase II Study of a Temozolomide-Based Chemoradiotherapy Regimen for High-Risk Low-Grade Gliomas
Brief Title: Temozolomide and Radiation Therapy in Treating Patients With Gliomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTOG 0424; CDR0000434849; NCI-2009-00723 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2005-06-13; First posted 2005-06-14 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2022-05

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult diffuse astrocytoma; adult oligodendroglioma; adult mixed glioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma; Oligodendroglioma; Glioma | interventions — Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Temozolomide + Radiation Therapy (RT) (Experimental): Daily temozolomide plus concurrent radiotherapy followed by temozolomide
  Interventions: Drug: Temozolomide; Radiation: Radiation therapy

INTERVENTIONS:
Drug: Temozolomide — Concurrent chemoradiotherapy temozolomide given 75 mg/m^2 daily during radiotherapy for 6 weeks.
  Post-Radiation Temozolomide given 150 mg/m2 daily on days 1-5 every 28 days with cycle one beginning 28 days post-radiotherapy. In the absence of grade 3 or 4 adverse events, a single dose escalation to 200 mg/m2/day could be attempted for cycle 2 and, if tolerated, that dose should continue for all subsequent cycles. Cycles were repeated every 28 days (+/- 2 days) for a total of 12 cycles.
Radiation: Radiation therapy — One treatment of 1.8 Gy given daily, 5 days per week (over 6 weeks) for a total dose of 54.0 Gy.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving temozolomide together with radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving temozolomide together with radiation therapy works in treating patients with low-grade gliomas.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the 3-year survival of patients with high-risk low-grade gliomas treated with temozolomide and radiotherapy followed by temozolomide alone with that of patients enrolled on European Organization for Research and Treatment of Cancer (EORTC)clinical trials EORTC-22844 and EORTC-22845.
* Determine the toxicity of this regimen in these patients.
* Determine the association between progression-free survival and O6-methylguanine-DNA methyltransferase (MGMT) methylation status in patients treated with this regimen.
* Determine the association between survival and MGMT methylation status in patients treated with this regimen.
* Determine the quality of life (QOL) of patients treated with this regimen.
* Determine the neurocognitive function of patients treated with this regimen.
* Evaluate the feasibility of collecting patient-reported QOL and neurocognitive assessments over 3 years.

OUTLINE: This is a non-randomized, multicenter study.

Patients receive oral temozolomide once daily on days 1-42 and undergo radiotherapy once daily on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36-40, one hour before RT weekdays, in the evening weekends. Beginning 28 days after completion of chemoradiotherapy, patients receive oral temozolomide once daily on days 1-5. Treatment with temozolomide repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, 6 months, 12 months.

After completion of study treatment, patients are followed at 4 months, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 135 patients will be accrued for this study within 44 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed* supratentorial glioma of 1 of the following histologies:

  * Astrocytoma (diffuse fibrillary, protoplasmic, or gemistocytic)
  * Oligodendroglioma
  * Oligoastrocytoma Note: *Histologic atypia allowed provided no other histologic features (i.e., frequent mitoses, endothelial proliferation, and/or acute necrosis) that would result in a designation of anaplastic astrocytoma, anaplastic mixed oligodendroglioma or oligoastrocytoma, or glioblastoma multiforme are present
* Unifocal or multifocal disease
* World Health Organization (WHO) grade II disease
* Neurofibromatosis allowed
* Surgical biopsy or resection for tumor tissue sampling required within the past 12 weeks

  * Tissue block or core biopsy available for O6-methylguanine-DNA methyltransferase analysis and tissue banking
  * Patients who have only had a stereotactic biopsy are not eligible
* Must have ≥ 3 of the following risk factors:

  * Age 40 and over
  * Largest preoperative tumor diameter ≥ 6 cm
  * Tumor crosses the midline
  * Astrocytoma-dominant tumor subtype
  * Preoperative Neurological Function Status > 1
* No other low-grade glioma histologies, including any of the following:

  * Pilocytic astrocytoma
  * Subependymal giant cell astrocytoma of tuberous sclerosis
  * Subependymoma
  * Pleomorphic xanthoastrocytoma
  * Presence of a neuronal element, such as ganglioglioma
  * Dysneuroembryoplastic epithelial tumor
* No high-grade glioma, including any of the following:

  * Anaplastic astrocytoma
  * Glioblastoma multiforme
  * Anaplastic oligodendroglioma
  * Anaplastic oligoastrocytoma
* No tumors in any non-supratentorial location, including any of the following:

  * Optic chiasm
  * Optic nerve(s)
  * Pons
  * Medulla
  * Cerebellum
  * Spinal cord
* No evidence of disease progression to spinal meninges or noncontiguous cranial meninges (i.e., leptomeningeal gliomatosis) by MRI of the spine or cerebrospinal fluid (CSF) cytology

  * MRI of the spine or CSF cytology are not required for patients without symptoms of spinal/cranial meningeal disease progression

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Total bilirubin ≤ 1.5 mg/dL
* Serum glutamate oxaloacetate transaminase (SGOT) or Serum glutamate pyruvate transaminase (SGPT) ≤ 2 times normal
* Alkaline phosphatase ≤ 2 times normal

Renal

* Serum creatinine ≤ 1.5 mg/dL

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known HIV positivity
* No other malignancy within the past 5 years except carcinoma in situ of the cervix or nonmelanoma skin cancer
* No active infection

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunotherapy or biologic therapy

Chemotherapy

* No prior chemotherapy
* No other concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy to the head and neck unless head and neck radiotherapy clearly excluded the brain (e.g., localized radiotherapy to the vocal cords)
* No prior radiotherapy to the brain
* No concurrent intensity modulated radiotherapy
* No concurrent stereotactic boost radiotherapy

Surgery

* See Disease Characteristics

Other

* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2005-01; Primary Completion 2013-02 (Actual); Study Completion 2022-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J. Fisher, MD, Principal Investigator — London Health Sciences Centre; David R. Macdonald, MD, FRCPC, Study Chair — London Health Sciences Centre; Glenn J. Lesser, MD, Study Chair — Wake Forest University Health Sciences; Stephen W. Coons, MD, Study Chair — St. Joseph's Hospital and Medical Center, Phoenix
Locations (47):
- United States (45):
  - Arizona Oncology Services Foundation, Phoenix, Arizona
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Integrated Community Oncology Network at Southside Cancer Center, Jacksonville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Baptist Medical Center South, Jacksonville, Florida
  - Integrated Community Oncology Network, Jacksonville Beach, Florida
  - Integrated Community Oncology Network - Orange Park, Orange Park, Florida
  - Florida Cancer Center - Palatka, Palatka, Florida
  - Flagler Cancer Center, Saint Augustine, Florida
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - DeCesaris Cancer Institute at Anne Arundel Medical Center, Annapolis, Maryland
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Kansas City, Kansas City, Missouri
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Cancer Research UK Medical Oncology Unit at Churchill Hospital & Weatherall Institute of Molecular Medicine - Oxford, Salem, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
- Canada (2):
  - Hopital Notre-Dame du CHUM, Montreal, Quebec
  - McGill Cancer Centre at McGill University, Montreal, Quebec

REFERENCES:
- [Derived] Bell EH, Zhang P, Fisher BJ, Macdonald DR, McElroy JP, Lesser GJ, Fleming J, Chakraborty AR, Liu Z, Becker AP, Fabian D, Aldape KD, Ashby LS, Werner-Wasik M, Walker EM, Bahary JP, Kwok Y, Yu HM, Laack NN, Schultz CJ, Gray HJ, Robins HI, Mehta MP, Chakravarti A. Association of MGMT Promoter Methylation Status With Survival Outcomes in Patients With High-Risk Glioma Treated With Radiotherapy and Temozolomide: An Analysis From the NRG Oncology/RTOG 0424 Trial. JAMA Oncol. 2018 Oct 1;4(10):1405-1409. doi: 10.1001/jamaoncol.2018.1977. PMID 29955793

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Temozolomide + Radiation Therapy (RT)
Started | 136
Completed | 129 (Subjects with data available for the primary analysis are considered to have completed the study.)
Not Completed | 7
Not completed — Protocol Violation | 7

BASELINE CHARACTERISTICS:
Population: Eligible patients
Arm/Group | Temozolomide + Radiation Therapy (RT)
Number analyzed (Participants) | 129
Age, Continuous [Median (Full Range); unit: years] | 49 [20 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 75

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival Rate at 3 Years
Description: Survival time is defined as time from registration to date of death from any cause and is estimated by the Kaplan-Meier method. Patients last known to be alive are censored at the date of last contact. This analysis was planned to occur when all patients had been potentially followed for at least 3 years.
Time Frame: Registration to 3 years
Population: Eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Temozolomide + Radiation Therapy (RT)
Number analyzed (Participants) | 129
percentage of participants | 73.1 [65.3 to 80.8]
Statistical Analysis 1: Comparison: Temozolomide + Radiation Therapy (RT); Assuming exponential distribution of survival times, the null hypothesis was a 43% increase in median survival time (40.5 mo. to 57.9 mo.) and a 21% increase in 3-year survival rate (54% to 65%). Assuming 5% ineligibility, 72 patients were required to be accrued over 3 years with 3-years of follow-up resulting in 80% power and 1-sided 0.10 significance level. (N later increased to 135 to accommodate an additional separate analysis of O-6-Methylguanine-DNA Methyltransferase (MGMT) status.); Test type: Superiority or Other; p < 0.001, Z-test

2. Primary Outcome: Progression-free Survival
Description: Progressive Disease (PD) is defined as 25% or > increase in the cross-sectional area of enhancing or non-enhancing tumor on consecutive MRI scans, or any new area(s) of tumor. Under exceptional circumstances, disease progression may be declared in the absence of an increase in tumor size based on "clinical deterioration" including the need for increasing doses of steroid and/or a worsening Karnofsky Performance Status(KPS) / Neurologic Function Score(NFS). Progression-free survival time is defined as time from registration to date of progressive disease or death from any cause and is estimated by the Kaplan-Meier method. Patients last known to be alive are censored at the date of last contact. Median survival time is reported.
Time Frame: From registration to last follow-up, up to 7.1 years. Analysis occurs after all patients have been on study for at least 3 years.
Population: Eligible patients
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Temozolomide + Radiation Therapy (RT)
Number analyzed (Participants) | 129
years | 4.5 [3.5 to NA] — Upper limit not reached

3. Primary Outcome: Survival and Progression-free Survival by O(6)-Methylguanine-DNA Methyltransferase (MGMT) Methylation Status
Description: Survival time is defined as time from registration to date of death from any cause. Progressive Disease (PD) is defined as 25% or > increase in the cross-sectional area of enhancing or non-enhancing tumor on consecutive MRI scans, or any new area(s) of tumor. Under exceptional circumstances, disease progression may be declared in the absence of an increase in tumor size based on "clinical deterioration" including the need for increasing doses of steroid and/or a worsening Karnofsky Performance Status(KPS) / Neurologic Function Score(NFS). Survival and progression-free survival are estimated by the Kaplan-Meier method. Patients last known to be alive are censored at the date of last contact.
Time Frame: Registration to 3 years
Population: Eligible patients with O(6)-methylguanine-DNA methyltransferase (MGMT) status
Measure: Median (95% Confidence Interval); unit: years
Groups:
- Temozolomide + Radiation Therapy (RT) - Methylated: Daily temozolomide plus concurrent radiotherapy followed by temozolomide - Patients with methylated status
- Temozolomide + Radiation Therapy (RT) - Unmethylated: Daily temozolomide plus concurrent radiotherapy followed by temozolomide - Patients with unmethylated status
Arm/Group | Temozolomide + Radiation Therapy (RT) - Methylated | Temozolomide + Radiation Therapy (RT) - Unmethylated
Number analyzed (Participants) | 57 | 18
years
  Overall Survival | NA [5.9 to NA] — Upper limit was not reached | 3.0 [2.3 to NA] — Upper limit was not reached
  Progression-free Survival | NA [4.5 to NA] — Median and upper limit were not reached | 2.0 [0.9 to 4.9]
Statistical Analysis 1: Comparison: Temozolomide + Radiation Therapy (RT) - Methylated vs Temozolomide + Radiation Therapy (RT) - Unmethylated; Overall survival: The sample size was increased to 135 to ensure adequate power to detect a hazard ratio (HR) of 2.5 for MGMT status, at a 2-sided significance level of 0.05 with an MGMT prevalence rate of at least 30%; Test type: Superiority; p = 0.0006, Log Rank — Two-sided significance level of 0.05; Hazard Ratio (HR) = 3.52, 95% CI 2-sided [1.64 to 7.56] — Reference level = Methylated
Statistical Analysis 2: Comparison: Temozolomide + Radiation Therapy (RT) - Methylated vs Temozolomide + Radiation Therapy (RT) - Unmethylated; Progression-free survival; Test type: Superiority; p = 0.0007, Log Rank — Two-sided significance level of 0.05; Hazard Ratio (HR) = 3.06, 95% CI 2-sided [1.55 to 6.04] — Reference level = Methylated

4. Primary Outcome: Quality of Life as Measured by the Functional Assessment of Cancer Therapy Scale With Brain Module (FACT-BR)
Description: Functional Assessment of Cancer Therapy Scale with brain module (FACT-BR): a 50-question self-report questionnaire contains the following domains (scales): Physical well-being (7 questions totalling 0-28), social/family well-being (7 questions totalling 0-28), emotional well-being (6 questions totalling 0-24), functional well-being (7 questions totalling 0-28) and brain cancer subscale which contains concerns relevant to patients with brain tumors (19 questions totalling 0-76). Each question has a value 0-4. For some questions a higher indicates better outcome and others are the opposite. The former are summed as is, the latter are reversed in value before adding, such that each domain ranges from 0 to 4 multiplied by the number of questions in the domain, with 0 indicating worst and the highest possible value indicating best outcome. The FACT-Br total (0-184) is obtained by adding all domains together if the overall question response rate is greater than 80%.
Time Frame: Baseline, 6 months, and 12 months.
Population: Eligible patients entered after QOL component amendment and alive at 6 and 12 months for respective post-baseline endpoints.
Measure: Median (Full Range); unit: units on a scale
Groups:
- Temozolomide + Radiation Therapy (RT) at Baseline; Temozolomide + Radiation Therapy (RT) at 6 Months; Temozolomide + Radiation Therapy (RT) at 12 Months: Daily temozolomide plus concurrent radiotherapy followed by temozolomide
Arm/Group | Temozolomide + Radiation Therapy (RT) at Baseline | Temozolomide + Radiation Therapy (RT) at 6 Months | Temozolomide + Radiation Therapy (RT) at 12 Months
Number analyzed (Participants) | 97 | 95 | 92
units on a scale
  Physical Well-Being: number analyzed (Participants) | 85 | 53 | 41
  Physical Well-Being | 23 [5.0 to 28.0] | 22 [3.0 to 28.0] | 23 [8.0 to 28.0]
  Social/Family Well-Being: number analyzed (Participants) | 81 | 50 | 40
  Social/Family Well-Being | 24.5 [7.0 to 28.0] | 24.0 [9.0 to 28.0] | 24.3 [8.0 to 28.0]
  Emotional Well-Being: number analyzed (Participants) | 86 | 54 | 42
  Emotional Well-Being | 18.5 [4.0 to 24.0] | 20.0 [11.0 to 24.0] | 23.0 [6.0 to 24.0]
  Functional Well-Being: number analyzed (Participants) | 86 | 54 | 42
  Functional Well-Being | 17.0 [2.0 to 28.0] | 18.0 [4.0 to 28.0] | 19.5 [2.0 to 28.0]
  Brain Cancer Subscale: number analyzed (Participants) | 86 | 55 | 43
  Brain Cancer Subscale | 54.0 [23.0 to 76.0] | 52.0 [22.0 to 75.0] | 59.0 [19.0 to 76.0]
  FACT-Br Total: number analyzed (Participants) | 80 | 50 | 40
  FACT-Br Total | 135.3 [69.5 to 184.0] | 129.9 [87.0 to 176.0] | 140.0 [65.0 to 181.0]

5. Primary Outcome: Neurocognitive Function
Description: Hopkins Verbal Learning Test (HVLT) is a test measuring learning memory retrieval, and memory consolidation processes.; Controlled Oral Word Association Test (COWAT) is a test of phonemic verbal fluency. The patient produces as many words as possible in 1 min. (each) for a specific letter (C, F, L or P, R, W).; Trail Making Test (TMT) is a measure of visuospatial scanning, attention, sequencing, and speed in Part A (TMT A) and executive function in Part B (TMT B). Patients must "connect the dots" either in a numbered sequence or alternating letters and numbers. Difference between pre-treatment baseline and follow-up assessment scores determined by the reliable change (RC) index, using a 90% confidence interval to designate statistically significant change.
Time Frame: Baseline, 6 months, and 12 months.
Population: Eligible patients entered after QOL component amendment with baseline score and alive at 6 and 12 months for respective timepoint.
Measure: Number; unit: participants
Arm/Group | Temozolomide + Radiation Therapy (RT) at 6 Months | Temozolomide + Radiation Therapy (RT) at 12 Months
Number analyzed (Participants) | 95 | 92
participants
  HVLT Recall Status: Deterioration: number analyzed (Participants) | 50 | 45
  HVLT Recall Status: Deterioration | 11 | 8
  HVLT Recall Status: No change: number analyzed (Participants) | 50 | 45
  HVLT Recall Status: No change | 26 | 22
  HVLT Recall Status: Improvement: number analyzed (Participants) | 50 | 45
  HVLT Recall Status: Improvement | 13 | 15
  COWA Status: Deterioration: number analyzed (Participants) | 49 | 43
  COWA Status: Deterioration | 1 | 3
  COWA Status: No change: number analyzed (Participants) | 49 | 43
  COWA Status: No change | 42 | 28
  COWA Status: Improvement: number analyzed (Participants) | 49 | 43
  COWA Status: Improvement | 6 | 12
  TMT A Status: Deterioration: number analyzed (Participants) | 50 | 45
  TMT A Status: Deterioration | 15 | 7
  TMT A Status: No change: number analyzed (Participants) | 50 | 45
  TMT A Status: No change | 24 | 24
  TMT A Status: Improvement: number analyzed (Participants) | 50 | 45
  TMT A Status: Improvement | 11 | 14
  TMT B Status: Deterioration: number analyzed (Participants) | 49 | 44
  TMT B Status: Deterioration | 11 | 7
  TMT B Status: No change: number analyzed (Participants) | 49 | 44
  TMT B Status: No change | 27 | 22
  TMT B Status: Improvement: number analyzed (Participants) | 49 | 44
  TMT B Status: Improvement | 11 | 15

ADVERSE EVENTS:
Description: Subjects experiencing more than one of a given adverse event are counted only once for that adverse event.
Arm/Group | Temozolomide + Radiation Therapy (RT)
Serious Adverse Events (participants affected / at risk) | 37/129
Other Adverse Events (participants affected / at risk) | 129/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Temozolomide + Radiation Therapy (RT) (N=129)
Blood/bone marrow - Other: (Blood and lymphatic system disorders) | 1
Atrial tachycardia (Cardiac disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 1
Dry eye NOS (Eye disorders) | 1
Abdominal pain NOS (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Small intestinal stricture NOS (Gastrointestinal disorders) | 1
Vomiting NOS (Gastrointestinal disorders) | 1
Disease progression NOS (General disorders) | 1
Fatigue (General disorders) | 6
Pain - Other: (General disorders) | 1
Hypersensitivity NOS (Immune system disorders) | 1
Infection - Other: (Infections and infestations) | 2
Infectous meningitis (Infections and infestations) | 1
Pneumonia NOS (Infections and infestations) | 1
Urinary tract infection NOS (Infections and infestations) | 1
Fracture NOS (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Leukopenia NOS (Investigations) | 2
Lymphopenia (Investigations) | 1
Neutrophil count (Investigations) | 3
Platelet count decreased (Investigations) | 8
Dehydration (Metabolism and nutrition disorders) | 2
Hyperglycaemia NOS (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Muscle weakness, generalized or specific area (not due to neuropathy): Extremity-lower (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Secondary Malignancy - possibly related to cancer treatment (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral ischaemia (Nervous system disorders) | 1
Cognitive disorder (Nervous system disorders) | 1
Convulsions NOS (Nervous system disorders) | 13
Depressed level of consciousness (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 2
Headache (Nervous system disorders) | 1
Hemorrhagic stroke (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 2
Personality change (Psychiatric disorders) | 1
Uterine hemorrhage (Reproductive system and breast disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dermatitis exfoliative NOS (Skin and subcutaneous tissue disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Hypertension NOS (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Temozolomide + Radiation Therapy (RT) (N=129)
Hemoglobin (Blood and lymphatic system disorders) | 53
Hearing impaired (Ear and labyrinth disorders) | 11
Ocular/visual - Other: (Eye disorders) | 8
Vision blurred (Eye disorders) | 10
Abdominal pain NOS (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 61
Diarrhoea NOS (Gastrointestinal disorders) | 27
Dry mouth (Gastrointestinal disorders) | 11
Dyspepsia (Gastrointestinal disorders) | 10
Gastrointestinal - Other: (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 96
Vomiting NOS (Gastrointestinal disorders) | 55
Edema: limb: (General disorders) | 7
Fatigue (General disorders) | 115
Pain - Other: (General disorders) | 9
Pyrexia (General disorders) | 8
Dermatitis radiation NOS (Injury, poisoning and procedural complications) | 36
Radiation recall syndrome (Injury, poisoning and procedural complications) | 10
Alanine aminotransferase increased (Investigations) | 38
Aspartate aminotransferase increased (Investigations) | 27
Blood alkaline phosphatase increased (Investigations) | 17
Blood creatinine increased (Investigations) | 12
Gamma-glutamyltransferase increased (Investigations) | 12
Leukopenia NOS (Investigations) | 67
Lymphopenia (Investigations) | 57
Metabolic/laboratory - Other: (Investigations) | 14
Neutrophil count (Investigations) | 35
Platelet count decreased (Investigations) | 58
Weight decreased (Investigations) | 28
Anorexia (Metabolism and nutrition disorders) | 57
Dehydration (Metabolism and nutrition disorders) | 9
Hypercalcaemia (Metabolism and nutrition disorders) | 7
Hyperglycaemia NOS (Metabolism and nutrition disorders) | 49
Hypernatremia (Metabolism and nutrition disorders) | 10
Hypoalbuminemia (Metabolism and nutrition disorders) | 13
Hypocalcemia (Metabolism and nutrition disorders) | 11
Hypoglycemia NOS (Metabolism and nutrition disorders) | 9
Hypokalemia (Metabolism and nutrition disorders) | 16
Hyponatremia (Metabolism and nutrition disorders) | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Muscle weakness, generalized or specific area (not due to neuropathy): Extremity-lower (Musculoskeletal and connective tissue disorders) | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 8
Ataxia (Nervous system disorders) | 10
Cognitive disorder (Nervous system disorders) | 16
Convulsions NOS (Nervous system disorders) | 45
Dizziness (Nervous system disorders) | 31
Dysgeusia (Nervous system disorders) | 32
Headache (Nervous system disorders) | 76
Memory impairment (Nervous system disorders) | 49
Neurology - Other: (Nervous system disorders) | 13
Peripheral motor neuropathy (Nervous system disorders) | 12
Peripheral sensory neuropathy (Nervous system disorders) | 25
Speech disorder (Nervous system disorders) | 14
Tremor (Nervous system disorders) | 14
Anxiety (Psychiatric disorders) | 16
Confusional state (Psychiatric disorders) | 13
Depression (Psychiatric disorders) | 20
Insomnia (Psychiatric disorders) | 34
Personality change (Psychiatric disorders) | 7
Pollakiuria (Renal and urinary disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 19
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12
Alopecia (Skin and subcutaneous tissue disorders) | 88
Dermatitis exfoliative NOS (Skin and subcutaneous tissue disorders) | 19
Dermatology/skin - Other: (Skin and subcutaneous tissue disorders) | 8
Pruritus (Skin and subcutaneous tissue disorders) | 10

LIMITATIONS AND CAVEATS:
Quality of life endpoint was added via an amendment while study was in progress.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes